CLINICAL TRIAL: NCT00088101
Title: Phase I Trial of STA-5312 Administered on Alternate Weekdays Every Two Weeks to Patients With Hematological Malignancies and Patients With Solid Tumors
Brief Title: STA-5312 Administered on Alternate Weekdays Every Two Weeks to Patients With Hematologic Malignancies and Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5312-01
Record Dates: First submitted 2004-07-20; First posted 2004-07-21 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Hematological Malignancies; Leukemia; Lymphoma; Metastatic or Unresectable Solid Tumors
Keywords: Hematological Malignancies; Leukemia; Lymphoma; Metastatic; Unresectable solid tumors
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia; Lymphoma; Neoplasm Metastasis

INTERVENTIONS:
Drug: STA-5312

SUMMARY:
The purpose of this study is to determine the safety, toxicity and patient tolerance of STA-5312 administered intravenously to patients with relapsed or refractory hematological malignancies and patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years or older with one of the following malignancies:
* Histologically or cytologically confirmed hematological malignancy (other than Acute Myeloid Leukemia and Myelodysplastic Syndrome) and if treatment is medically indicated, or,
* Histologically-confirmed non-hematological malignancy that is metastatic or unresectable and for which no standard therapy is available.
* Patients with CLL, PLL, CML, CTCL, ATL, and Non-Hodgkin's Lymphoma may be entered if they are refractory to or have relapsed following conventional chemotherapy regimens such as alkylating agents (e.g. chlorambucil and cyclophosphamide), anthracycline combinations [e.g. CHOP (cyclophosphamide, doxorubicin, vincristine, prednisone)], and/or purine analogues (e.g. fludarabine monophosphate and 2-CDA) and are not currently being considered for re-treatment with conventional regimens
* Patients with CLL and other leukemic malignancies will be staged according to the modified Rai staging criteria [low-risk, intermediate-risk and high risk]. All patients in the high-risk group (Stage III and IV) are eligible. Intermediate risk patients (Stage I and II) with one or more criteria of active disease (such as progressive lymphocytosis, lymphadenopathy, and splenomegaly, weight loss > 10% within 6 months, extreme fatigue, fever and/or night sweats without evidence of infection, etc.) are also eligible
* ECOG Performance Status of 0-2
* Life expectancy of greater than 12 weeks.
* Patients must have acceptable organ and marrow function at screening and pre-dose visits as defined below unless approved medically by the clinical investigator.
* Absolute neutrophils count greater than 1,000 cells/ul for patients with hematologic malignancies and ≥1,500 cells/ul for patients with solid tumors
* Platelets greater than 100,000/ul
* Hgb greater than 8.5 g/dL
* Total bilirubin must be <1.5 mg/dL or < 2X upper limit of normal
* AST (SGOT) < 2.5 times the upper limit of normal
* ALT (SGPT) < 2.5 times the upper limit of normal
* Adequate renal function (serum creatinine < 2.0 mg/dL or a calculated creatinine clearance greater than 50 mL/min)
* Electrocardiogram without evidence of clinically significant conduction abnormalities or active ischemia as determined by the investigator.
* NCI grade 0-1 left ventricular ejection fraction within 30 days of dosing.
* The effects of STA-5312 on the developing human fetus are unknown. Therefore, women of childbearing potential (defined as women under 50 years of age or history of amenorrhea for < 12 months prior to study entry) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform the treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Women who are pregnant or lactating.
* Patients who have had chemotherapy, radiotherapy (except palliative radiation delivered to < 20% of bone marrow), immunotherapy, or corticosteroids ( > 10 mg/day of prednisone or equivalent) within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* The use of nitrosoureas or mitomycin C within 6 weeks prior to study entry.
* Patients with prior peripheral blood stem cell rescue or bone marrow transplantation.
* History of primary brain tumors or active brain metastases. (Patients with previously treated brain metastases who are not receiving corticosteroids or anticonvulsants may be considered for enrollment)
* History of stroke or other significant neurologic limitations within 6 months prior to study enrollment
* Use of any investigational agents within 4 weeks of study enrollment.
* History of severe allergic reactions to excipients (e.g. Tween 80) or had hypersensitivity reactions to other chemotherapeutic agents similar in structure to STA-5312.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, as determined by the investigator.
* History of active CNS-lymphoma, AIDS-related lymphoma, or any uncontrolled severe medical illness or infection.
* Grade 2 or higher sensory or motor neuropathy at screening.
* Major surgery (excluding that for diagnosis) within 4 weeks of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2004-02; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Wilshire Oncology Medical Group, Pomona, California
  - Baptist Cancer Institute, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Tufts New England Medical Center, Boston, Massachusetts
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Carolinas HealthCare System, Charlotte, North Carolina
  - The West Clinic, Memphis, Tennessee
  - The Sarah Cannon Cancer Center, Nashville, Tennessee